CLINICAL TRIAL: NCT00013403
Title: The Impact of Rehabilitation on Quality of Life in Visually Impaired
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1998R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Blindness
Keywords: Vision, quality of life
MeSH Terms: conditions — Blindness

INTERVENTIONS:
Procedure: Blindness

SUMMARY:
The project has four primary objectives: 1) Determine if blind rehabilitation improves the quality of life of legally blind veterans; 2) Determine the relationship between quality of life and visual function; 3) Determine if factors, such as cognitive status, level of depression, age and the presence of additional medical conditions besides vision loss, intervention of blind rehabilitation extends beyond the visually impaired individual and improve the quality of life of their primary caregiver (e.g. spouse, partner, family member or friend.)

ELIGIBILITY:
Visually impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1999-04; Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Birmingham, Birmingham, Alabama, United States